CLINICAL TRIAL: NCT05452005
Title: Fluorine-18-AlphaVBeta6-Binding Peptide Positron Emission Tomography for Staging, Response Assessment, and Patient Selection in Metastatic Non-Small Cell Lung Cancer
Brief Title: Fluorine-18-AlphaVBeta6-Binding Peptide Positron Emission Tomography in Metastatic Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Julie L. Sutcliffe, Ph.D, Professor of Internal Medicine and Biomedical Engineering, University of California, Davis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1718953
Record Dates: First submitted 2022-06-28; First posted 2022-07-11 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer; Lung Cancer Metastatic; Brain Metastases; Non Small Cell Lung Cancer
Keywords: Positron Emission Tomography
MeSH Terms: conditions — Lung Neoplasms; Brain Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental [18F]-αvβ6-BP (Experimental): Patients receive [18F]-αvβ6-BP BP IV and then undergo a PET/CT scan over 30 minutes 60 minutes post-injection.
  Interventions: Drug: [18F]-αvβ6-BP

INTERVENTIONS:
Drug: [18F]-αvβ6-BP — Subjects will be injected twice with up to 10 millicurie (mCi) of 18F-αvβ6-BP as a rapid intravenous (i.v) bolus.

SUMMARY:
This study investigates fluorine-18-AlphaVBeta6-BP ([18F]-αvβ6-BP) as a Positron Emission (PET) imaging agent in Non-Small Cell Lung Cancer (NSCLC) patients with brain metastases. Investigators hypothesize that [18F]-αvβ6-BP PET/Computed Tomography (CT) is a sensitive tool for disease assessment in patients with metastatic NSCLC, including those with brain metastases.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

The primary objective of this study is to evaluate the sensitivity and specificity of [18F]-αvβ6-BP PET/CT for detecting metastases in patients with NSCLC.

OUTLINE:

Patients will undergo [18F]-αvβ6-BP PET/CT at baseline in addition to standard-of-care [18F]-2-fluoro-2-deoxy-D-glucose (FDG) PET/CT body and magnetic resonance imaging (MRI) of the brain. Patients will then undergo standard-of-care cancer directed therapy. Patients will be re-staged 8-12 weeks later at the next standard-of-care imaging time point with [18F]-αvβ6-BP PET/CT, [18F]-FDG PET/CT, and MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age >18 yrs
2. Biopsy proven NSCLC with brain metastases (treated or untreated)
3. Life-expectancy of ≥3 months in the opinion of the treating physician
4. Available archival tumor tissue (excisional, core, or fine needle aspiration (FNA) is acceptable). Tissue from a metastatic site is preferred when available.
5. Able to tolerate all study procedures, including remain motionless for up to 30-60 minutes per scan
6. Ability to understand and willingness to sign a written informed consent document.
7. Planned to undergo additional cancer-directed therapy followed by standard-of-care re-staging imaging
8. [18F]-FDG PET/CT within 21 days of enrollment
9. MRI brain within 21 days of enrollment
10. Eastern Cooperative Oncology Group Performance Status ≤ 2
11. Glomerular filtration rate (GFR) ≥ 60

Exclusion Criteria:

1. Pregnant or lactating women
2. Prisoners
3. Concurrent malignancy of a different histology that could confound imaging interpretation
4. Patients who cannot undergo PET/CT scanning because of weight limits(>350lbs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
[18F]-αvβ6-BP PET/CT imaging compared to immunohistochemistry | Up to six months
  Standard uptake value (SUV) values from [18F]-αvβ6-BP PET/CT will be compared to immunohistochemistry (IHC) αvβ6 staining of archival tissue to assess the sensitivity of [18F]-αvβ6-BP PET/CT to detect αvβ6 positive metastasis in NSCLC

SECONDARY OUTCOMES:
Comparison of standard-of-care MRI and [18F]-αvβ6-BP PET/CT imaging | Up to six months
  Detection of lesions with [18F]-αvβ6-BP will be compared to the number of lesions identified during standard-of-care MRI imaging
Comparison of standard-of-care [18F]-FDG PET/CT and [18F]-αvβ6-BP PET/CT imaging | Up to six months
  SUVmax values obtained during standard-of-care FDG/PET will be compared to SUVmax values obtained from [18F]-αvβ6-BP PET/CT imaging
Comparison of standard-of-care MRI brain and [18F]-FDG PET/CT and [18F]-αvβ6-BP PET/CT imaging post treatment | Up to six months
  Lesion response will be assessed based on standard-of-care MRI images, [18F]-FDG PET/CT and [18F]-αvβ6-BP PET/CT post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Julie L. Sutcliffe, PhD, Principal Investigator — The Regents of the University of California (Davis)
Locations (1):
- The University of California Davis Comprehensive Cancer Center, Sacramento, California, United States